CLINICAL TRIAL: NCT06842953
Title: Is an Adjustment in the Recommended Indoor Temperature Upper Limit of 26°C Required During Higher Levels of Humidity?
Brief Title: Influence of Indoor Humidity on Physiological Strain in Older Adults During a Simulated Heat Wave
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ottawa (Other)
Responsible Party: Principal Investigator, Glen P. Kenny, Full Professor, University of Ottawa
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: HEPRU-2025-02-A
Record Dates: First submitted 2025-02-17; First posted 2025-02-24 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Heat Stress; Physiological Stress
Keywords: Heat wave; Indoor overheating; Thermoregulation; Heat strain; Elderly; Heat vulnerability; Hyperthermia; Thermal comfort
MeSH Terms: conditions — Heat Stress Disorders; Hyperthermia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Exposure to recommended indoor temperature limit with normal indoor humidity (Experimental): Participants exposed daylong (10 hours) to an indoor temperature maintained at 26°C and 45% relative humidity (humidex equivalent of 29).
  Interventions: Other: Simulated indoor overheating
- Exposure to recommended indoor temperature limit with low indoor humidity (Experimental): Participants exposed daylong (10 hours) to an indoor temperature maintained at 26°C and 15% relative humidity (humidex equivalent of 23).
  Interventions: Other: Simulated indoor overheating
- Exposure to recommended indoor temperature limit with high indoor humidity (Experimental): Participants exposed daylong (10 hours) to an indoor temperature maintained at 26°C and 85% relative humidity (humidex equivalent of 37).
  Interventions: Other: Simulated indoor overheating
- Exposure to high indoor temperature with normal indoor humidity (Experimental): Participants exposed daylong (10 hours) to an indoor temperature maintained at 31°C and 45% relative humidity (humidex equivalent of 37).
  Interventions: Other: Simulated indoor overheating

INTERVENTIONS:
Other: Simulated indoor overheating — Older adults are exposed to a 10-hour simulated exposure

SUMMARY:
Laboratory-based studies show that exposure to high humidity can worsen the effects of heat stress in young and older adults by impeding sweat evaporation - the main mechanism by which the human body cools itself. At high levels of humidity, the efficiency of sweating decreases causing a greater rise core temperature and burden on the cardiovascular system. In this context, increasing temperatures and humidity with climate change thus pose a potential compound risk for human health. While humidity's role in heat-health outcomes could substantially alter projections of health burdens from climate change, the impact of humidity on physiological strain in vulnerable people in relation to the indoor environment has yet to be evaluated. In a recent study delineating the physiological effects of the proposed 26°C indoor upper limit (PMID: 38329752), relative humidity was set to 45% in all conditions based on indoor humidity standards by the American Society of Heating and Air-Conditioning Engineers. However, it is unknown whether a refinement of the recommended indoor temperature limit of 26°C is required in situations where humidity cannot be maintained at this level.

On separate occasions, the investigators will assess the change in body temperature and cardiovascular strain in older adults (65-85 years) exposed for 10 hours at the recommended indoor temperature limit of 26°C and 45% relative humidity (equivalent humidex of 29 (considered comfortable)) (experimental condition A), to 26°C with a relative humidity of 15% (equivalent humidex of 23 (considered comfortable); humidex is used to measure the perceived temperature taking into account the humidity)) (experimental condition B), to 26°C with a relative humidity of 85% (equivalent humidex of 37 (considered somewhat uncomfortable)) (experimental condition C), and to 31°C and 45% relative humidity with an equivalent humidex of 37 (considered somewhat uncomfortable) that is similar to experimental condition C. With this experimental design, investigators will assess the effects of indoor humidity in driving human heat strain and identify whether refinements in the recommended 26°C indoor temperature limit may be required. Further, by evaluating changes in relation to ambient conditions with a similar humidex, the investigators can assess how individuals perceive and respond to both heat and humidity.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking.
* English or French speaking.
* Ability to provide informed consent.
* with or without a) chronic hypertension (elevated resting blood pressure; as defined by Heart and Stroke Canada and Hypertension Canada), b) type 2 diabetes as defined by Diabetes Canada, with at least 5 years having elapsed since time of diagnosis

Exclusion Criteria:

* Episode(s) of severe hypoglycemia (requiring the assistance of another person) within the previous year, or inability to sense hypoglycemia (hypoglycemia unawareness).
* Serious complications related to diabetes (gastroparesis, renal disease, uncontrolled hypertension, severe autonomic neuropathy).
* Uncontrolled hypertension - BP >150 mmHg systolic or >95 mmHg diastolic in a sitting position.
* Restrictions in physical activity due to disease (e.g. intermittent claudication, renal impairment, active proliferative retinopathy, unstable cardiac or pulmonary disease, disabling stroke, severe arthritis, etc.).
* Use of or changes in medication judged by the patient or investigators to make participation in this study inadvisable.
* Cardiac abnormalities identified during screening

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-03-14 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Core temperature (Peak) during daylong exposure to indoor overheating | End of 10 hour daylong exposure
  Peak rectal temperature (15 min average) during exposure. Rectal temperature is measured continuously throughout the 10 hours of the simulated indoor overheating.
Core temperature (AUC) during daylong exposure to indoor overheating | End of 10 hour daylong exposure
  Areas under the curve (AUC) of rectal temperature during the 10 hour simulate indoor overheating.
Heat rate (Peak) during daylong exposure to indoor overheating | End of 10 hour daylong exposure
  Peak heart rate (15 min average) during exposure. Heart rate is measured continuously throughout the 10 hours of the simulated indoor overheating.
Heart rate (AUC) during daylong exposure to indoor overheating | End of 10 hour daylong exposure
  Areas under the curve (AUC) of heart rate during the 10 hour simulate indoor overheating.
Cardiac response to standing from supine (30:15 Ratio) during daylong exposure to indoor overheating | At the start (hour 0) and end of 10 hour daylong exposure
  Cardiac response to standing evaluated as the ratio between the highest R-wave to R-wave interval (lowest heart rate) measured at the 30th heart beat after standing from supine (+/- 5 beats) and the lowest R-wave to R-wave interval (highest heart rate) measured at the 15th heart beat after standing (+/- 5 beats). Cardiac response to standing will be evaluated twice, during two lying-to-standing tests (separated by 10 min of supine rest).
Systolic Response to Standing From Supine during daylong exposure to indoor overheating | At the start (hour 0) and end of 10 hour daylong exposure
  Systolic blood pressure response to standing evaluated as the difference in blood pressure measured between the standing and supine. Standing systolic blood pressure will be taken as the lowest value of those measured after 60 and 120 seconds of standing. Systolic response to standing will be evaluated twice, during two lying-to-standing tests (separated by 10 min of supine rest).
Heart rate variability: RMSSD during daylong exposure to indoor overheating | At the start (hour 0) and end of 10 hour daylong exposure
  Root mean squared standard deviation of normal-to-normal R-wave to R-wave intervals (RMSSD) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the supine position. RMSSD will be evaluated twice, during two paced breathing periods (separated by 4 min of supine rest).
Heart rate variability: SDNN during daylong exposure to indoor overheating | At the start (hour 0) and end of 10 hour daylong exposure
  Standard deviation of normal-to-normal R-wave to R-wave intervals (SDNN) measured during 5 minutes of paced breathing (15 breaths/min) with participants in the supine position. SDNN will be evaluated twice, during two paced breathing periods (separated by 4 min of supine rest).
Thermal comfort scale during daylong exposure to indoor overheating | At the start (hour 0) and end of 10 hour daylong exposure
  Thermal comfort assessed via a visual analog scale ranging from extremely uncomfortable to extremely comfortable (midpoint: neutral).
Thirst sensation scale during daylong exposure to indoor overheating | At the start (hour 0) and end of 10 hour daylong exposure
  Thermal sensation assessed via a visual analog scale ranging from extremely hot to neutral (midpoint: hot).
Arousal scale during daylong exposure to indoor overheating | At the start (hour 0) and end of 10 hour daylong exposure
  Felt arousal scale assessed via a visual analog scale ("How worked up are you?") ranging from "high arousal" to "low arousal".
Fluid loss during daylong exposure to indoor overheating | At end of 10 hour daylong exposure
  Average hourly fluid consumption calculated by weighing participant water intake at the start and end of each hour of exposure (normalized to the exposure duration).
Changes in plasma volume during daylong exposure to indoor overheating | At end of 10 hour daylong exposur
  Change in plasma volume from baseline values calculated from duplicate measurements of hemoglobin and hematocrit at the start and end of each exposure using the technique by Dill and Costill
Systolic blood pressure during daylong exposure to indoor overheating | At the start (hour 0) and end of 10 hour daylong exposure
  Systolic blood pressure measured in triplicate via automated oscillometry (~60 seconds between measures)
Rate pressure product during daylong exposure to indoor overheating | At the start (hour 0) and end of 10 hour daylong exposure
  Rate pressure product, an index of myocardial work and strain, calculated as systolic blood pressure x heart rate.

SECONDARY OUTCOMES:
Impulse control (cognitive function) during daylong exposure to indoor overheating | At the start (hour 0) and end of 10 hour daylong exposure
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of impulse control. Participants will be asked to respond to both "go" and "no-go" visual cues. In response to the "go" cue, participants will initiate a movement of the device.
Memory recall (cognitive function) during daylong exposure to indoor overheating | At the start (hour 0) and end of 10 hour daylong exposure
  Participants will be provided with a tablet device with the Sway Medical testing platform for the assessment of memory recall. Participants complete both a delayed recall test and a working memory test.
CDC 4-Stage Balance Test (Postural stability) during daylong exposure to indoor overheating | At the start (hour 0) and end of 10 hour daylong exposure
  To assess postural stability, participants hold a tablet to their chest, then auditory cues guide participants through four consecutive stances, feet side by side, instep of one foot touching the big toe of the other foot, tandem stand with one foot in front of the other, heel touching toe, and stand on one foot. The balance assessment will be evaluated based on movement detected by an accelerometer integrated into the hardware of the tablet device (Sway Medical Inc).
BTrackS Balance Assessment (Postural stability) during daylong exposure to indoor overheating | At the start (hour 0) and end of 10 hour daylong exposure
  To assess postural stability, participants will be asked to stand on a BTracks force plate with their feet spread out to shoulder width, hand on their hips and eyes closed. The assessment will comprise of four trials (one practice trial) lasting 20 seconds in length and 20 seconds between trials. Center of pressure (COP) vector data along vertical (y) and horizontal (x) axes will be summed for the total path excursion length (cm) during each trial.
Profiles of Mood States (POMS) during daylong exposure to indoor overheating | At the start (hour 0) and end of 10 hour daylong exposure
  Potential changes in mood (7 subscales of mood: tension, anger, depression, fatigue, confusion, vigor and esteem-related affect). The POMS-40 is a validated, self-administered questionnaire that examines seven distinct aspects of mood state across two positive subscales (Esteem-Related Affect, and Vigor) and five negative subscales (Fatigue, Tension, Confusion, Anger, and Depression), which are described across 40 distinct adjectives (reference). For each individual item, participants were asked to describe "how you feel right now" by responding using a 5-point Likert scale (0 = "Not at all", 1 = "A little", 2 = "Moderately", 3 = "Quite a lot", or 4 = "Extremely"). The values of items associated with a specific subscale (e.g., Fatigue) were summed to calculate its score.
Environmental Symptoms Questionnaire (ESQ) during daylong exposure to indoor overheating | At the start (hour 0) and end of 10 hour daylong exposure
  Self-reported environmental reactions and medical symptomatology associated with prolonged heat exposure. The ESQ-IV is a validated 68-item, self-administered questionnaire that has been used successfully in identifying symptomatology during exposure to a wide variety of environmental conditions, including heat exposure [24, 25]. Participants are asked to assess and described "how you have been feeling today" by responding to each item using a 6-point Likert scale (0 = "Not at all", 1 = "Slight", 2 = "Somewhat", 3 = "Moderate", 4 = "Quite a bit", or 5 = "Extreme"). Total Symptom Score was calculated from this data by taking the sum of the intensity ratings from all 68 individual items using reverse scores for the three positive items from the list ("I Felt Good", "I Felt Alert", and "I Felt Wide Awake").
Sleepiness during daylong exposure to indoor overheating A | At the start (hour 0) and end of 10 hour daylong exposure
  Karolinska sleepiness scale measures the subjective level of sleepiness at a particular time
Sleepiness during daylong exposure to indoor overheating B | At the start (hour 0) and end of 10 hour daylong exposure
  Stanford sleepiness scale consists of only one item, where participant must identify one of seven statements that best represents their level of perceived sleepiness. It employs a scale of 1 to 7 with 1 = feeling wide awake and 7 = sleep onset soon

CONTACTS AND LOCATIONS:
Locations (1):
- University of Ottawa, Ottawa, Ontario, Canada